CLINICAL TRIAL: NCT00682812
Title: Significance of the High-risk Hpv Viral Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2007-A01335-48; 2007-30
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: HPV Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 125 womens with normal cervix
  Interventions: Other: 2 cervical takings and 2 sampling of blood
- 2 (Other): 105 womens with an intraepithelial lesion
  Interventions: Other: 2 cervical takings and 2 sampling of blood
- 3 (Other): 105 womens with a cancer of the cervix
  Interventions: Other: 2 cervical takings and 2 sampling of blood

INTERVENTIONS:
Other: 2 cervical takings and 2 sampling of blood — * 2 cervical takings
  * 2 sampling of blood before and after the total hysterectomy
  Arms: 1
Other: 2 cervical takings and 2 sampling of blood — * cervical taking during the cervical conization
  * 2 sampling of blood before and after the intervention
  Arms: 2
Other: 2 cervical takings and 2 sampling of blood — * cervical taking during the pelvien examination under general anesthetic realized systematically during the balance sheet of pre-therapeutic evaluation
  * 2 sampling of blood before and after the intervention
  Arms: 3

SUMMARY:
The aim of this study is to evaluate the significance of an elevated high-risk HPV (HR-HPV) viral load.

DETAILED DESCRIPTION:
We will particularly evaluate if the HR-HPV viral load:

* Is correlated to the transcription of the genes of the oncoproteins E6 and E7
* Is predictive of the integration of the virus in infected cells
* Is predictive of the presence of HPV in patients' blood
* Influences the local and systemic immunologic response

ELIGIBILITY:
Inclusion Criteria:

* The women consulting for the therapeutic care (by hysterectomy or conization) of a LIEHG or a cervical cancer (carcinoma epidermoid or adenocarcinoma) confirmed by the anatomopathologique analysis of a preoperative cervical biopsy.
* The women having a normal cervix consulting for the surgical care by hysterectomy of a good-hearted pathology of the womb. The normality of the cervix will be confirmed by the anatomopathologique analysis of the detail of hysterectomy
* The patients participating in this study will have to be of more than 18 years old. All the subjects will be profitable of a regime of Social Security.

Exclusion Criteria:

* The patients having a LIEBG
* The patients incapable to receive the information enlightened on the progress and the objectives of the study
* The patients not having signed enlightened assent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2008-06-16 (Actual); Primary Completion 2014-04-24 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Estimate the meaning of a viral load raised in HPV oncogenic | 36 months

SECONDARY OUTCOMES:
To estimate the correlation enters the vorale load of the HPV oncogenic and the severity of the cervical hurt | 36 months
Estimate the correlation between the viral load of the HPV oncogenic and the level of transcription of the genes coding for oncoproteines E6 and E7 | 36 months
Estimate the correlation between the viral load in HPV oncogenic and the integration of the viral genome in that of the infected cells | 36 months
Estimate the correlation between a viral load raised in HPV oncogenic and a presence of HPV in the circulating blood of the infected patients | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Xavier CARCOPINO, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Hopital Nord, service de gynécologie-obstétrique, Marseille, France